CLINICAL TRIAL: NCT02199587
Title: The Effect of Medical Clown on the Pain and Anxiety Perception During LRH Analog Treatment or Growth Hormone Provocation Test
Brief Title: The Effect of Medical Clown on the Pain and Anxiety Perception During LRH Analog Treatment or GH Provocation Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MeirMc069-14CTIL
Record Dates: First submitted 2014-06-18; First posted 2014-07-24 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Precocious Puberty; Growth Hormone Tests
Keywords: Medical clown; Growth hormone; Precocious puberty
MeSH Terms: conditions — Puberty, Precocious

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endocrine test with medical clown (Active Comparator): children who are referred to endocrine test will have the procedure with a medical clown, or without. The pain and anxiety perception of the child and caregivers will be compare between the two scenarios
  Interventions: Behavioral: Presence of medical clown during endocrine test
- Endocrine test without medical clown (No Intervention)

INTERVENTIONS:
Behavioral: Presence of medical clown during endocrine test
  Arms: Endocrine test with medical clown

SUMMARY:
The investigators would like to examine the contribution of medical clowns in routine medical procedures in the endocrine clinic. This will be the first time that will objective evaluate the effect of medical clown on stress hormone such as adrenaline cortisol and prolactin, and also evaluate the effect of mental stress on growth hormone secretion in children.

The aim of the current study is testing the pain and anxiety of the patient and the accompanying parent and medical staff in the presence or absence of medical clown at the time:

1. LRH analog (decapeptyl) intramuscular injections for precocious puberty.
2. Growth hormone tests.

Secondary end point will be:

1. Changes in stress hormones: cortisol , prolactin and adrenalin during growth hormone tests in the presence of a clown.
2. Does the presence of a medical clown and the mental stress affect the secretion of growth hormone?
3. Are there differences in growth hormone secretion and stress hormones between the various tests for growth hormone secretion (glucagon, clonidine or arginine) in the presence of a clown?
4. Are there differences in response to stress and the secretion of growth hormone in children with obesity?

DETAILED DESCRIPTION:
80 children from the endocrine clinic who are referred for treatment with LRH analog or directed to growth hormone tests, will take part in the study:

1.40 children who are referred to decapeptyl treatment will receive the injection once with a medical clown, and the next time with out the clown and vise verse. The pain and anxiety perception of the child and caregivers will be compare between the two scenarios. The children will be randomly assigned to begin treatment in the presence of a clown and the next injection without medical clown and the second group starts the injections without medical clown and the next shot in the presence of a clown.

2.40 children from endocrine clinic who are referred for growth hormone tests because of short stature will have the test with or without medical clown in a random selection.

Procedure

1. Children who receive decapeptyl injections once a month. Before getting the shot will be offered to participate in the study. After signing the consent form and parent consent they randomized to get the treatment in the presence of a clown or without health.
2. The kids and their parents who referred to growth hormone test will be offered to participate in the study and after signing the consent will be invited for the test. According to accepted protocol, the children arrived after overnight fast, an intravenous line is inserted and blood is taken for measurement of human growth hormone levels, IGF1, thyroid function test, prolactin, cortisol, and adrenaline and then a stimulates substance (glucagon, clonidine or arginine) is given. Afterward blood tests for human growth hormone and cortisol levels, are taken every 30-60 minutes for approximately 3-4 hours after administration of the provocative substance. During the test regular vital signs are monitored according to Protocol.

In both procedures, anxiety of the child and his parent will be evaluated by questionnaires. State-Trait (STAI) Inventory questionnaires for the parent and STAIC questionnaires for the kids. In addition, the kid, his parent and the medical staff will evaluate for pain by Visual Analog Score (VAS).

Inclusion criteria:

* Children older than 4 years.
* referred by the endocrine clinic to a decapeptyl treatment or growth hormone test.

The criteria included:

• The consent of a parent and the child to participate in a study

Questionnaires Anxious parent questionnaire (STAI). Anxiety questionnaire (STAIC)

Pain assessment scale:

Pain assessment by the child, the parents and the staff (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Children older than 4 years. referred by the endocrine clinic to a decapeptyl treatment or growth hormone test.

Exclusion Criteria:

* none

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2014-12-17 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
change from base line of the anxiety of the child and his parent by State-Trait (STAI) Inventory questionnaires for the parent and STAIC questionnaires for the kids. | At 30 min before the procedure and 30 min after the procedure

SECONDARY OUTCOMES:
Changes in hormones: cortisol , Growth hormone, prolactin and adrenalin during growth hormone tests in the presence of a clown. | At 30 min before the test and 30 min after the test

CONTACTS AND LOCATIONS:
Overall Officials: nitsan dror, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center endocrine unit, Kfar Saba, Israel